CLINICAL TRIAL: NCT05869422
Title: Randomised, Double-blind, Placebo-controlled Clinical Trial Evaluating the Effectiveness of a Low-dose Iron Supplementation in Non-anaemic Iron-deficient Women
Brief Title: Low-dose Iron Supplementation in Non-anaemic Iron-deficient Women
Acronym: PCLDIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Krayenbühl GmbH (Industry)
Responsible Party: Principal Investigator, Albina Nowak, PD Dr. med., University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LowDoseIronVsPlacebo; SNCTP000005680 (Registry Identifier: Swiss National Clinical Trial Portal (SNCTP))
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Iron Deficiency (Without Anemia)
Keywords: iron deficiency; low dose iron therapy; iron therapy
MeSH Terms: conditions — Iron Deficiencies | interventions — Iron

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: study employees
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): placebo tablet containing no iron
  Interventions: Other: Placebo
- Low Dose Iron (Experimental): low-dose tablet containing 6mg of iron
  Interventions: Dietary Supplement: Iron

INTERVENTIONS:
Dietary Supplement: Iron — 60 ± 5 days of daily oral iron supplementation.
  Arms: Low Dose Iron
Other: Placebo — 60 ± 5 days of daily oral placebo intake.
  Arms: Placebo

SUMMARY:
The goal of this study is to investigate the efficacy of a low dose iron supplement (6mg) compared to a placebo tablet.

DETAILED DESCRIPTION:
The established therapy for iron-deficiency today is oral iron supplementation. However, this often leads to side effects such as constipation, black stools, nausea, and abdominal pain. There are some studies that have compared the efficacy of low-dose iron with normal-dose iron. These showed that the side effects are dose-dependent. Furthermore, some studies have shown that the uptake capacity of high-dose iron is less efficient due to the upregulation of hepcidin. In a pilot study with low-dose iron (6mg per tablet), a significant increase in iron was shown, which can be explained by a lower hepcidin release. Therefore, the investigators would like to show the efficacy of the low-dose iron product in a placebo-controlled setting. Furthermore, the goal is to examine the reduction of side effects before and after administration of the iron and placebo tablet. Additionally, a potential increase of low blood pressure to normal blood pressure will be investigated. There will be two groups of women: one group will be given a low-dose iron supplement of two tablets containing each 6mg for 2 months (60 days), the other one will get two placebo tablet for 2 months, accordingly.

ELIGIBILITY:
Inclusion Criteria:

* informed consent as documented by signature
* female gender
* premenopausal
* age > 18 years
* regular menstrual cycle
* BMI in normal range (18-25 kg/m²)
* serum-ferritin ≤30µg/l
* no anaemia (Hemoglobin ≥117g/l)
* no intake of dietary supplements containing iron (last 4 weeks)
* the participant is linguistically and cognitively able to understand the study procedure

Exclusion Criteria:

* Current pregnancy
* breastfeeding
* hypermenorrhea (more than 5 unties/tampons per day)
* chronic inflammatory diseases (e.g. colitis)
* psychiatric disorders
* chronic kidney disease (creatinine >80 µmol/l)
* liver disease (ALT >35 U/l)
* increased CRP (>5mg/l)
* hypersensitivity to iron-supplements
* intake of medicines that interact with oral iron supplementation (e.g. PPI)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 59 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Serum-ferritin change | 60 ± 5 days
  significant change of serum-ferritin under supplementation

SECONDARY OUTCOMES:
Blood Pressure | 60 ± 5 days
  change of blood pressure (systolic and diastolic blood pressure)
Blood Sugar | 60 ± 5 days
  change of blood sugar levels
Lipid Status | 60 ± 5 days
  change of lipid status (total cholesterol, HDL, LDL, triglycerides)

OTHER OUTCOMES:
Safety Endpoint | 60 ± 5 days
  Incidence of adverse events during 2 months under low dose iron supplementation and placebo treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided